CLINICAL TRIAL: NCT07325097
Title: A Prospective, Single Arm Study to Assess the Safety and Tolerability of PVEK Corneal Implant for the Treatment of Corneal Edema
Brief Title: PVEK Corneal Implant For Treatment of Corneal Edema
Acronym: CIFRE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Precise Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-CRN-001
Record Dates: First submitted 2025-12-22; First posted 2026-01-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Corneal Edema; Fuchs' Endothelial Dystrophy; Pseudophakic Bullous Keratopathy; Corneal Endothelial Dysfunction
Keywords: Endothelial keratoplasty; Tissue-engineered corneal implant; Corneal endothelial cells; Collagen scaffold
MeSH Terms: conditions — Corneal Edema; Fuchs' Endothelial Dystrophy | interventions — Drug Implants

STUDY DESIGN:
Intervention Model Description: PVEK
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PVEK (Experimental): Participants undergo implantation of the PVEK tissue-engineered corneal endothelial implant in a single administration
  Interventions: Combination Product: Precise Vision Endothelial Keratoplasty (PVEK) Implant

INTERVENTIONS:
Combination Product: Precise Vision Endothelial Keratoplasty (PVEK) Implant — PVEK is a tissue-engineered corneal endothelial implant intended to treat corneal endothelial dysfunction. The implant consists of a human collagen scaffold (support layer) and corneal endothelial cells (drug substance). The product is pre-loaded in a sterile injector/cartridge system that serves as the packaging and transplantation device and is ready for use. It is shipped in corneal storage media and is delivered into the anterior chamber during endothelial keratoplasty.

SUMMARY:
The goal of this clinical trial is to learn if PVEK, a corneal implant , is safe and well tolerated for people with corneal swelling caused by Fuchs' endothelial dystrophy or pseudophakic bullous keratopathy who need endothelial keratoplasty.

The main questions it aims to answer are:

What side effects may happen after the PVEK implant?

How many participants can complete the first 6 months after surgery without needing another treatment because the implant did not help enough or was not tolerable?

This is a Phase 1 (first-in-human) study with one study group, meaning all participants receive the PVEK implant (there is no placebo or comparison group). About 15 participants will take part and will be followed for up to 12 months after surgery.

Participants will:

Complete screening tests (including eye exams and routine health checks)

Have the PVEK implantation surgery

Use prescribed eye drops after surgery

Return for follow-up visits over the next 12 months for eye exams and tests (such as vision testing, eye pressure checks, and eye scans)

ELIGIBILITY:
Inclusion Criteria:

age 18/50 years or older

Corneal edema requiring endothelial keratoplasty due to Fuchs' endothelial dystrophy and/or pseudophakic bullous keratopathy

Pseudophakic study eye

Best corrected visual acuity (BCVA) in the study eye between 6/379 (1.8 logMAR) and 6/12 (0.3 logMAR)

Central corneal thickness greater than 0.6 mm by OCT

Exclusion Criteria:

Phakic study eye

Study eye is a "single sight eye" (per protocol definition) / fellow eye does not meet protocol vision requirement

Malpositioned intraocular lens (dislocation/subluxation) in the study eye

Prior ocular procedure in the study eye other than uncomplicated cataract surgery with a stable, centered posterior chamber IOL

Axial length below 21 mm or above 26 mm

Other significant corneal disease (beyond mild dry eye) or prior keratoplasty in the study eye, or visually significant corneal scarring/opacities not expected to improve with treatment

Active ocular or eyelid infection/inflammation; active/prior herpetic ocular infection; uveitis

Glaucoma / history or suspicion of elevated IOP, or screening IOP above 23 mmHg (either eye)

Synechiae; abnormal anterior segment (e.g., aphakia, aniridia)

Corneal endothelial cell density above 1000 cells/mm² at screening (or not reliably measurable)

Uncontrolled systemic conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and treatment-emergent adverse events (TEAEs) | 6 months
  Number and percentage of participants with any adverse event (AE) and any treatment-emergent adverse event (TEAE) occurring after PVEK implantation.
Proportion of participants completing 6-month follow-up without seeking alternative treatment | 6 months
  Percentage of participants who complete the 6-month follow-up without seeking alternative treatment due to perceived lack of efficacy or intolerability of side effects.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) from 6 to 12 months after PVEK implantation | 6-12 months
  Number and percentage of participants with any adverse event (AE) .
Elevated IOP | 12 months
  Number and percentage of participants with increased intraocular pressure (IOP) greater than 26 mmHg
BCVA | 12 months
  change from baseline in best corrected visual acuity (BCVA)
Central corneal thickness | 12 months
  Central corneal thickness measurements by OCT
Corneal endothelial cell density | 6 and 12 months
  Corneal endothelial cell density assessed by specular microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Minouni, Prof., Principal Investigator — Rambam Health Care Campus
Locations (3):
- Ophthalmological Center After S.V.Malayan, Yerevan, Armenia
- Israel (2):
  - Sharei Zedek Medical Center, Jerusalem, Jerusalem
  - Rambam Medical Center, Haifa

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available to other researchers